CLINICAL TRIAL: NCT02593201
Title: The Efficacy of Prolonged Antibiotic Therapy for the Prevention of Relapsing Peritonitis in Peritoneal Dialysis Patients With High Dialysis Effluent Bacterial DNA Fragment Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPDNA
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Peritoneal Dialysis
MeSH Terms: interventions — Cefazolin; Ceftazidime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): One extra week of antibiotic therapy
  Interventions: Drug: Extended antibiotics (cefazolin or ceftazidime)
- Control (Sham Comparator): No extra antibiotics
  Interventions: Drug: Usual antibiotics (cefazolin or ceftazidime)

INTERVENTIONS:
Drug: Extended antibiotics (cefazolin or ceftazidime) — To continue with the existing effective antibiotic therapy for one extra week
  Arms: Treatment
Drug: Usual antibiotics (cefazolin or ceftazidime) — Usual duration of effective antibiotic therapy therapy
  Arms: Control

SUMMARY:
Peritoneal dialysis (PD) is the first-line treatment of end stage renal disease (ESRD) in Hong Kong. Despite the advances in antibiotic therapy and connecting system, recurrent peritonitis remains the major cause of peritoneal failure. A recent study showed that an elevated bacterial DNA fragment levels in PD effluent 5 days prior to the completion of antibiotics predicts the development of relapsing or recurrent peritonitis episodes. We hypothesize that prolonged antibiotic therapy in PD patients with peritonitis and high PD effluent bacterial DNA fragment levels could prevent the development of relapsing and recurrent peritonitis. We plan to conduct a randomized control study of 360 patients with PD peritonitis. After inform consent, they will be randomized to receive one additional week of the effective antibiotic treatment (the Preemptive Treatment Group) or no additional treatment (the Control Group). Specimens of PD effluent will be collected 5 days prior to the completion of antibiotics for the measurement of bacterial DNA fragments. All patients will be followed for 6 months after completion of antibiotic therapy for the development of relapsing, recurrent, or repeat peritonitis episodes. Our study will determine the efficacy of a test-before-treat algorithm that could reduce the incidence of relapsing and recurrent peritonitis and, at the same time, minimize the unnecessary use of prolonged antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peritoneal dialysis-related peritonitis

Exclusion Criteria:

* Patients with fungal peritonitis
* Patients with obvious surgical problems and require laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
relapsing peritonitis episodes | 6 months
repeat peritonitis episodes | 6 months
recurrent peritonitis episodes | 6 months

SECONDARY OUTCOMES:
peritonitis that requires hospitalization | 6 months
need of catheter removal | 6 months
  by record review
need of conversion to long-term hemodialysis | 6 months
  by record review
death due to peritonitis | 6 months
all cause mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong